CLINICAL TRIAL: NCT04249895
Title: Comprehensive Digital Archive of Cancer Imaging-Radiation Oncology( CHAVI-RO )
Status: Completed | Type: Observational
Sponsor: Tata Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: EC/GOVT/24/IRB23
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: All Cancer
Keywords: Carcinoma; Radiomics; Image Processing; Radiology; Molecular Biology; Data Analytics Center; Artificial Intelligence; Medical Physics; Big Data; Radiation Oncology
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main Cohort: All patients are undergoing radiotherapy in Tata Medical Center

SUMMARY:
In this pilot project Investigators propose to create annotated image data bank of patients suffering from cancer. The system will provide India's first comprehensive platform to upload annotated images with associated medical and demographic information of a patient. It will support flexible query from the users with appropriate choice from a set of attributes and design of various query filters using a GUI. Over the proposed period of 18 months, images and records related to radiation oncology including pretreatment images of at least 500 patients would be annotated and archived in the data bank. The imaging modalities to be covered are X-RAY mammograms, SPECT, CT, CBCT, MR, PET-CT, Ultrasound, digital histopathology, etc. In this phase, this study will include data sets of five types of cancers namely, breast, head and neck, brain, cervix and lung cancer.

Investigator propose to demonstrate the application of this data set in cancer research. Investigator will work on serial PET-CT based radiomics of breast and cervix cancer patients to extract appropriate features and correlate them with clinico-pathological variants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing radiotherapy planned with volumetric imaging.

-

Exclusion Criteria:

* Informed Consent not given

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Patients undergoing radiotherapy in the dept of radiotherapy, Tata Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with complete data safe. | 18 months
  Count of patients with complete radiological, pathological and demographic information in the CHAVI RO database.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanjoy Chatterjee, Kolkata, West Bengal, India

IPD SHARING:
Plan to Share IPD: No